CLINICAL TRIAL: NCT02883426
Title: Evaluation of the Safety and Immunogenicity of Live Influenza A Vaccine H3N2v (6-2) AA ca Recombinant (A/Minnesota/11/2010 (H3N2v) x A/Ann Arbor/6/60 ca), a Live Attenuated Virus Vaccine Candidate for Prevention of Influenza H3N2v Disease
Brief Title: Evaluating the Safety and Immunogenicity of a Live Attenuated Virus Vaccine to Prevent Influenza H3N2v Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: URMC 16-001
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: H3N2v Influenza Viruses
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group 1: H3N2v Seronegative Adults: H3N2v LAIV (Experimental): Participants will receive one dose of H3N2v LAIV on Day 0 (study entry). They will then receive one dose of H3N2v IIV on Day 84.
  Interventions: Biological: H3N2v MN 2010/AA ca live attenuated influenza vaccine (LAIV); Biological: H3N2v inactivated subvirion influenza vaccine
- Group 2: H3N2v Seropositive Adolescents: H3N2v LAIV (Experimental): Participants will receive two doses of H3N2v LAIV, the first dose on Day 0 (study entry) and the second dose on Day 28. They will then receive one dose of H3N2v IIV on Day 84.
  Interventions: Biological: H3N2v MN 2010/AA ca live attenuated influenza vaccine (LAIV); Biological: H3N2v inactivated subvirion influenza vaccine
- Group 2: H3N2v Seropositive Adolescents: Placebo (Placebo Comparator): Participants will receive two doses of placebo, the first dose on Day 0 (study entry) and the second dose on Day 28. They will then receive one dose of H3N2v IIV on Day 84.
  Interventions: Biological: H3N2v inactivated subvirion influenza vaccine; Biological: Placebo
- Group 3: H3N2v Seronegative Adolescents: H3N2v LAIV (Experimental): Participants will receive two doses of H3N2v LAIV, the first dose on Day 0 (study entry) and the second dose on Day 28. They will then receive one dose of H3N2v IIV on Day 84.
  Interventions: Biological: H3N2v MN 2010/AA ca live attenuated influenza vaccine (LAIV); Biological: H3N2v inactivated subvirion influenza vaccine
- Group 3: H3N2v Seronegative Adolescents: Placebo (Placebo Comparator): Participants will receive two doses of placebo, the first dose on Day 0 (study entry) and the second dose on Day 28. They will then receive one dose of H3N2v IIV on Day 84.
  Interventions: Biological: H3N2v inactivated subvirion influenza vaccine; Biological: Placebo
- Group 4: Children: H3N2v LAIV (Experimental): Participants will receive two doses of H3N2v LAIV, the first dose on Day 0 (study entry) and the second dose on Day 28. They will then receive one dose of H3N2v IIV on Day 84.
  Interventions: Biological: H3N2v MN 2010/AA ca live attenuated influenza vaccine (LAIV); Biological: H3N2v inactivated subvirion influenza vaccine
- Group 4: Children: Placebo (Placebo Comparator): Participants will receive two doses of placebo, the first dose on Day 0 (study entry) and the second dose on Day 28. They will then receive one dose of H3N2v IIV on Day 84.
  Interventions: Biological: H3N2v inactivated subvirion influenza vaccine; Biological: Placebo

INTERVENTIONS:
Biological: H3N2v MN 2010/AA ca live attenuated influenza vaccine (LAIV) — Approximately 10^7.0 Fluorescent Focus Units (FFU) per 0.2 mL dose; administered intranasally
  Other Names: H3N2v LAIV
  Arms: Group 1: H3N2v Seronegative Adults: H3N2v LAIV; Group 2: H3N2v Seropositive Adolescents: H3N2v LAIV; Group 3: H3N2v Seronegative Adolescents: H3N2v LAIV; Group 4: Children: H3N2v LAIV
Biological: H3N2v inactivated subvirion influenza vaccine — 15 μg; administered intramuscularly
  Other Names: H3N2v IIV
Biological: Placebo — Administered by nasal spray
  Arms: Group 2: H3N2v Seropositive Adolescents: Placebo; Group 3: H3N2v Seronegative Adolescents: Placebo; Group 4: Children: Placebo

SUMMARY:
This study will evaluate the safety and immunogenicity of the H3N2v MN 2010/AA ca live attenuated influenza vaccine (H3N2v LAIV) in healthy children and adults, 6 to 26 years old.

DETAILED DESCRIPTION:
The potential for widespread human disease due to the H3N2v influenza viruses is considerable. Infection with these viruses would most likely impact young children. This study will evaluate the safety and immunogenicity of the H3N2v MN 2010/AA ca live attenuated influenza vaccine (H3N2v LAIV) in healthy children and adults, 6 to 26 years old.

The study will enroll participants sequentially in four groups: Group 1 will include H3N2v seronegative adults ages 18-26 years; Group 2 will include H3N2v seropositive adolescents ages 13-17 years; Group 3 will include H3N2v seronegative adolescents ages 13-17 years; and Group 4 will include children ages 6 to 12 years, who will not be screened for H3N2v serostatus.

At study entry (Day 0), participants in Group 1 will receive one dose of H3N2v LAIV. Participants in Groups 2, 3, and 4 will be randomly assigned to receive two doses of either H3N2v LAIV or placebo, receiving the first dose on Day 0 and the second dose on Day 28. On Day 84, all participants will receive one dose of H3N2v IIV (an inactivated booster vaccine).

Participants will attend several additional study visits through Day 180. These visits may include a physical examination; respiratory examination; and collection of blood, urine, or nasal fluids.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females between 6 and 26 years of age inclusive.
* For children, presence of an adult caregiver who is in good health and able to understand and carry out the requirements
* General good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator.
* Agree to storage of blood specimens for future research.
* Available for the duration of the trial.
* Willingness to participate in the study as evidenced by signing the informed consent document. Verbal assent will be obtained from minors 6 to 12 years of age and signed assent will be obtained from minors 13 and older.
* Female subjects of childbearing potential must agree to use effective birth control methods for the duration of the study (e.g., pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; intrauterine device; abstinence from heterosexual intercourse, surgical sterilization).

Exclusion Criteria:

* Anticipated direct routine [e.g. weekly or more frequent] contact with individuals younger than the designated age groups being studied as a result of household contact, occupation, or participation in day care with such individuals.
* Pregnancy as determined by a positive urine or serum human choriogonadotropin (β-HCG) test.
* Currently breast-feeding.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history or physical examination.
* Behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, affects the ability of the subject to understand and cooperate with the study protocol.
* Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
* History of anaphylaxis.
* Allergy to oseltamivir as determined by subject report.
* Current diagnosis of asthma or reactive airway disease (within the past 2 years).
* Use of aspirin or salicylate-containing medications within 28 days prior to randomization or expected receipt through 28 days after final vaccination.
* History of Guillain-Barré Syndrome.
* Known history of HIV, hepatitis C, or active hepatitis B infection.
* Known immunodeficiency syndrome.
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to vaccination.
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination.
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination.
* Travel to the Southern Hemisphere within 14 days prior to study vaccination.
* Travel on a cruise ship within 14 days prior to study vaccination.
* Receipt of another investigational vaccine or drug within 30 days prior to study vaccination.
* Allergy to eggs or egg products, gentamicin, or gelatin.
* Chronic use of intranasal medications.

Ages: 6 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events (REs) that occur during the acute monitoring phase of the study | Measured through Day 180
Area under the curve of nasal virus shedding after each dose of vaccine | Measured through Day 180
  As assessed by liquid titration of nasal secretions on Madin Darby canine kidney (MDCK) cells at 33°C
Development of serum antibody | Measured through Day 180
  Assessed by either hemagglutination inhibition (HAI) or microneutralization (MN) assays

SECONDARY OUTCOMES:
Development of a significant increase in nasal secretion hemagglutinin (HA)-specific antibody | Measured through Day 180
  Assessed by enzyme-linked immunosorbent assay (ELISA), luminex or microneutralization assay

CONTACTS AND LOCATIONS:
Overall Officials: John Treanor, M.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center (URMC), Vaccine Research Unit (Outpatient), Rochester, New York, United States